CLINICAL TRIAL: NCT02185950
Title: The Effects of Therapeutic Resources on Structure and Function of Normal and Burned Skin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Elaine Caldeira de Oliveira Guirro, Professor, PT, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1146-7342
Record Dates: First submitted 2013-08-15; First posted 2014-07-10 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-07

CONDITIONS: Burn; Skin Graft
Keywords: Burn; Skin graft; Elasticity; Skin; Physical therapy modalities
MeSH Terms: conditions — Burns | interventions — Ultrasonography; Paraffin Embedding

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Ultrasound group (Experimental): Therapeutic ultrasound, 3 MHz, continuous with intensity 1W/cm2 will be applied to the selected region (burn scar deep 2nd degree or 3rd degree, grafted) with exposure time of 2 minutes for each effective radiation area head (ERA), a total of 4 minutes of application in an area of 9X5 cm, and the application parameters with a matched control side of the patient, in a region with contralateral uninjured skin.
  Interventions: Device: ultrasound
- Group paraffin (Experimental): Paraffin therapy is heated with thermostat own equipment, being applied to the selected region (burn scar deep 2nd degree or 3rd degree, grafted) and control (uninjured), with a length of 9X5 cm, at a temperature of 38 ° C with appropriate brush in layers (4 layers), remaining for 20 minutes. After the period of application of paraffin will be removed and discarded, with no reuse.
  Interventions: Device: paraffin
- Ultrasound group + endermotherapy (Experimental): Therapeutic ultrasound, 3 MHz, continuous with intensity 1W/cm2 will be applied to the selected region (burn scar deep 2nd degree or 3rd degree, grafted) with exposure time of 2 minutes for each effective radiation area head (ERA), a total of 4 minutes of application in an area of 9X5 cm. The application of endermotherapy will be held shortly after the therapeutic ultrasound in a timely manner across the surface of the scar, for about 2 seconds per head area with a negative pressure between 100-200 mmHg, a total of 4 minutes application in an area of 9 x 5 cm. The same application parameters will be performed with one hand matched control patient, in a region with contralateral uninjured skin.
  Interventions: Device: ultrasound; Device: endermotherapy
- Group paraffin + endermotherapy (Experimental): Paraffin therapy is heated with thermostat own equipment, being applied to the selected region (burn scar deep 2nd degree or 3rd degree, grafted) and control (uninjured), with a length of 9X5 cm, at a temperature of 38 ° C with appropriate brush in layers (4 layers), remaining for 20 minutes. After the period of application of paraffin will be removed and discarded, with no reuse.The application of endermotherapy will be held shortly after the paraffin therapy in a timely manner across the surface of the scar, for about 2 seconds per head area with a negative pressure between 100-200 mmHg, a total of 4 minutes application in an area of 9 x 5 cm. The same application parameters will be performed with one hand matched control patient, in a region with contralateral uninjured skin.
  Interventions: Device: paraffin; Device: endermotherapy

INTERVENTIONS:
Device: ultrasound
  Arms: Ultrasound group; Ultrasound group + endermotherapy
Device: paraffin
  Arms: Group paraffin; Group paraffin + endermotherapy
Device: endermotherapy
  Arms: Group paraffin + endermotherapy; Ultrasound group + endermotherapy

SUMMARY:
Burning produces changes in the biomechanical properties of the skin causing limitation of movement. The increase in skin suppleness is very important in the rehabilitation process, since its increase makes therapeutic interventions aimed at increasing the range of motion, thus improving functional pattern. Will be evaluated 60 volunteers of both sexes aged 20-80 years seen at the Burns Unit of the Clinical Hospital of the Faculty of Medicine of Ribeirão Preto. There will be a traditional physical therapy evaluation as well as evaluation of the specific characteristics of the burn and scar. The temperature of the region will be assessed by thermography, and biophysical parameters and biomechanical skin evaluated by Cutometer and their accessory probes (mexameter, reviscometer, sebometer) before, immediately after and 10, 20 and 30 minutes of application of therapeutic resources. Volunteers will undergo continuous application of ultrasound with 3 MHz and intensity of 1 W/cm2 in the region due to scar deep second degree burn or third degree, and the application time of 2 minutes for each effective radiation area of the head (ERA) in a predetermined region of 9X5 cm a total of 4 minutes of application, therapy paraffin 20 minutes and 4 minutes endermology negative pressure between 100 and 200mmHg, in a continuous mode with glass head (1.5cm in diameter .) Applications will be set by random draw (design crusader cross-over) with an interval of 7 days between applications (wash-out). The data will be submitted to analysis of normality by the Shapiro-Wilk test, and the behavior of the effect between groups and pre-and post-intervention will be evaluated by two-way ANOVA followed by post-hoc (Bonferroni) or Friedman, p <0.05

ELIGIBILITY:
Inclusion Criteria:

* Victims of deep second degree burns and third degree with a length of at least 1% of body surface area burned
* Postoperative graft skin (4 and 6 months)
* Anywhere in the body that has area to uninjured contralateral control
* Good state of physical and mental health
* Aged between 20 and 80 years
* Both genders
* Irrespective of race, class or social group

Exclusion Criteria:

* Volunteers with illnesses or deformities that may interfere with evaluation and procedures
* Volunteers which do not accept signing the Instrument of Consent and do not meet the inclusion criteria

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-06; Primary Completion 2015-01 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Elasticity of skin and scar | 3 years
  The measurement of skin and scar elasticity will be measured by the used a noninvasive assessment equipment, Cutometer.

SECONDARY OUTCOMES:
Erythema of skin and scar | 3 years
  The measurement of skin and scar erythema will be measured by the probe accessory Cutometer, Mexameter.
Fiber direction of skin and scar | 3 years
  The measurement of skin and scar fiber direction will be measured by the probe accessory Cutometer, Reviscometer.

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Guirro, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- University of São Paulo, RibeirãoPreto, São Paulo, Brazil

REFERENCES:
- See also: Related Info — http://www.fmrp.usp.br